CLINICAL TRIAL: NCT02505672
Title: Vestibular Function After Chemoradiotherapy for Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, yotam shkedy, Resident, Rabin Medical Center
Other Study IDs: 0361-14-RMC
Record Dates: First submitted 2015-07-18; First posted 2015-07-22 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Vestibular function; chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients older than 18 who are planned to undergo chemoradiotherapy for nasopharyngeal carcinoma.
  Interventions: Radiation: Chemoradiotherapy for nasopharyngeal carcinoma

INTERVENTIONS:
Radiation: Chemoradiotherapy for nasopharyngeal carcinoma — Note that this is standard care for NPC and patients are not assigned to different intervention groups. All patients in the study will receive the same treatment (chemoradiotherapy) and will be observed for changes in vestibular function.

SUMMARY:
Nasopharyngeal carcinoma (NPC) is usually treated with chemoradiotherapy. While the effects of this treatment on cochlear function is well characterized, its effect on vestibular function is not well studied.

In this study the investigators will study the vestibular function of 50 patients undergoing chemoradiotherapy for NPC both before and after treatment in order to better define its effects. All patients will undergo a validated questionnaire (dizziness handicap index), posturography, audiometry and vestibular-evoked myogenic potentials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Biopsy-proven NPC.
* About to undergo chemoradiotherapy with intensity-modulated radiotherapy (IMRT).

Exclusion Criteria:

* Pregnancy.
* Prior vestibular dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven nasopharyngeal carcinoma who are planned to undergo chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Subjective dizziness and vestibular dysfunction using the dizziness handicap index | 6 months after completion of treatment
Hearing level using standard audiometry | 6 months after completion of treatment
Objective vestibular function using posturography | 6 months after completion of treatment
Vestibular saccular function using vestibular-evoked myogenic potentials | 6 months after completion of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology, Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Colaco RJ, Betts G, Donne A, Swindell R, Yap BK, Sykes AJ, Slevin NJ, Homer JJ, Lee LW. Nasopharyngeal carcinoma: a retrospective review of demographics, treatment and patient outcome in a single centre. Clin Oncol (R Coll Radiol). 2013 Mar;25(3):171-7. doi: 10.1016/j.clon.2012.10.006. Epub 2013 Jan 18. PMID 23337060
- [Background] Tuan JK, Ha TC, Ong WS, Siow TR, Tham IW, Yap SP, Tan TW, Chua ET, Fong KW, Wee JT. Late toxicities after conventional radiation therapy alone for nasopharyngeal carcinoma. Radiother Oncol. 2012 Sep;104(3):305-11. doi: 10.1016/j.radonc.2011.12.028. Epub 2012 Jan 24. PMID 22280806
- [Background] Zhang L, Chen QY, Liu H, Tang LQ, Mai HQ. Emerging treatment options for nasopharyngeal carcinoma. Drug Des Devel Ther. 2013;7:37-52. doi: 10.2147/DDDT.S30753. Epub 2013 Feb 1. PMID 23403548
- [Background] Wei Y, Zhou T, Zhu J, Zhang Y, Sun M, Ding X, Wang D, Li H, Li B. Long-term outcome of sensorineural hearing loss in nasopharyngeal carcinoma patients: comparison between treatment with radiotherapy alone and chemoradiotherapy. Cell Biochem Biophys. 2014 Jul;69(3):433-7. doi: 10.1007/s12013-014-9814-x. PMID 24510513
- [Background] Lin C, Lin SW, Weng SF, Lin YS. Risk of developing sudden sensorineural hearing loss in patients with nasopharyngeal carcinoma: a population-based cohort study. Head Neck. 2014 Feb;36(2):203-8. doi: 10.1002/hed.23278. Epub 2013 Jun 18. PMID 23780872
- [Background] Tsang RK, Kwong DL, Ho AC, To VS, Ho WK, Wei WI. Long-term hearing results and otological complications of nasopharyngeal carcinoma patients: comparison between treatment with conventional two-dimensional radiotherapy and intensity-modulated radiotherapy. ORL J Otorhinolaryngol Relat Spec. 2012;74(4):228-33. doi: 10.1159/000341096. Epub 2012 Aug 17. PMID 22907195
- [Background] Chao WY, Tseng HZ, Tsai ST. Caloric response and postural control in patients with nasopharyngeal carcinoma after radiotherapy. Clin Otolaryngol Allied Sci. 1998 Oct;23(5):439-41. doi: 10.1046/j.1365-2273.1998.00170.x. PMID 9800080
- [Background] Chen PR, Hsu LP, Tu CE, Young YH. Radiation-induced oscillopsia in nasopharyngeal carcinoma patients. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):466-70. doi: 10.1016/j.ijrobp.2004.05.016. PMID 15667968
- [Background] Wu CC, Young YH, Ko JY. Effect of irradiation on vestibular evoked myogenic potentials in nasopharyngeal carcinoma survivors. Head Neck. 2003 Jun;25(6):482-7. doi: 10.1002/hed.10215. PMID 12784240
- [Background] Young YH, Ko JY, Sheen TS. Postirradiation vertigo in nasopharyngeal carcinoma survivors. Otol Neurotol. 2004 May;25(3):366-70. doi: 10.1097/00129492-200405000-00027. PMID 15129119
- [Background] Hsin CH, Chen TH, Young YH, Liu WS. Comparison of otologic complications between intensity-modulated and two-dimensional radiotherapies in nasopharyngeal carcinoma patients. Otolaryngol Head Neck Surg. 2010 Nov;143(5):662-8. doi: 10.1016/j.otohns.2010.07.012. PMID 20974336
- [Background] Kaplan DM, Friger M, Racover NK, Peleg A, Kraus M, Puterman M. [The Hebrew dizziness handicap inventory]. Harefuah. 2010 Nov;149(11):697-700, 750, 749. Hebrew. PMID 21250408